CLINICAL TRIAL: NCT03795103
Title: Effect of a Neuromuscular Electrical Stimulation Program on Walking Capacity in Peripheral Artery Disease Patients: a Randomized Controlled Trial
Brief Title: Effect of a Neuromuscular Electrical Stimulation Program on Walking Capacity in Peripheral Artery Disease Patients
Acronym: ELECTROPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: AD REM TECHNOLOGY (Unknown); Ecole Normale Supérieure de Rennes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35RC15_8961_ELECTROPAD
Record Dates: First submitted 2018-11-09; First posted 2019-01-07 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Arteriopathy
Keywords: Lower Extremity Peripheral Arterial Disease
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators won't know which arm is allocated to arteriopathic patients. Program will be send to patients by a outcome research engineer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients achieving neuromuscular electrical stimulation (Experimental): LEPAD patients achieving a 12-week program of neuromuscular electrical stimulation. Group of arteriopathic patients who will perform electrostimulation sessions at home and independently. These patients will also receive a study participation guide that will include an information leaflet outlining tips for active living and walking.
  Interventions: Device: neuromuscular electrical stimulator
- Control (Other): Group of artriopathic patients who will maintain their usual drug management. These patients will also receive a study participation guide that will include an information leaflet outlining tips for active living and walking.
  Interventions: Other: Advices
- Healthy volunteers (Other): Ancillary study. Participants will perform a precise program of walking sessions performed outdoors and independently and the same biological parameters as those assessed in arteriopathic patients will be assessed
  Interventions: Other: Walking sessions

INTERVENTIONS:
Device: neuromuscular electrical stimulator — A 12-week program of neuromuscular electrical stimulation
  Arms: Patients achieving neuromuscular electrical stimulation
Other: Walking sessions — A 12-week program of walking sessions performed outdoors and independently
  Arms: Healthy volunteers
Other: Advices — The usual practice associated with an information leaflet outlining tips for active living and walking.
  Arms: Control

SUMMARY:
Lower extremity peripheral arterial disease (LEPAD) is a highly prevalent chronic disease. Cardiovascular mortality of LEPAD patients at five years ranges between 18 to 30%. LEPAD is primarily caused by atherosclerosis that induces an inadequate blood flow to meet the tissues demand due to the narrowing of the arteries. An aggravation of the arterial lesions in LEPAD patients induces a worsening of patients' symptoms and a severe limitation of their walking capacity, contributing to an impairment of their quality of life.

Interventions designed to improve walking impairment may have a significant impact on the functional capacity in LEPAD patients. Lower extremity electrical stimulation is an older technique that relies on different types of electrical stimulations with different expected physiological effects on hemodynamics, skeletal muscle functions or pain pathway. The aim of the ELECTRO-PAD study is to assess the effect of a 12 weeks program of neuromuscular electrical stimulation (NMES) on the absolute walking distance (AWD) measured during a treadmill test in peripheral artery disease patients.

DETAILED DESCRIPTION:
The aim of the ELECTRO-PAD study is to assess the effect of a 12 weeks program of neuromuscular electrical stimulation (NMES) on the absolute walking distance (AWD) measured during a treadmill test in peripheral artery disease patients.

Arteriopatic patients will be randomized in 2 groups :

* patients submitted to a 12 weeks program of neuromuscular electrical stimulation (NMES group)
* patients without any program (control group) All patients will also receive a study participation guide that will include an information leaflet outlining tips for active living and walking.

After eligibility criteria will be assessed, patient will be included and randomized (visit 1). A second visit will be performed after 12 weeks (visit 2).

In parallel, 2 ancillary studies will be performed :

* Among Rennes' arteriopatic patients, endothelial function will be assessed using measures from 40 patients. Assessment will be done between 1 and 14 days after visit 1 (visit 1')
* The second ancillary study concerns 40 volunteers with no cardiac or vascular pathology, only in the coordinating center Rennes. The same measures will be performed for these volunteers and for arteriopatic patients.

ELIGIBILITY:
Inclusion Criteria:

Arteriopatic patients :

* Age > 40 years old.
* Subjects with Lower Extremity Peripheral Artery disease (LEPAD). LEPAD is defined by the presence of at least one of the following criteria:

  * History of revascularization in the lower limbs due to LEPAD; OR
  * Ankle brachial index (ABI) of ≤ 0.90; OR
  * ABI or ankle systolic blood pressure decrease during recovery from treadmill walking test > 20 % or > 30 mmHg, respectively; OR
  * Toe-brachial index ≤0.70 if ABI cannot be measured and if incompressible arteries are suspected.
* Complain of exertional calf pain (fatigue, discomfort or cramping) that can begin or not at rest, causes the participant to stop walking and relieves or lessens within 10 minutes of rest (assessed using the San Diego questionnaire AND confirmed during treadmill testing);
* Pain (fatigue, discomfort or cramping) is mainly located at the calves' level.
* Maximal walking distance on treadmill < 300 m (treadmill protocol 3.2 km/h, 10% grade);
* Subject receiving from at least one month the recommend medical therapy for LEPAD management (antiplatelet therapy and statin medication).
* Obtained informed consent.

Healthy volunteers

* Age > 50 years old;
* Absence of pain reported in the lower limbs during walking as supported by a negative score in the San Diego Questionnaire;
* Absence of any functional limitation during the treadmill walking test: 15 min of walking at 3.2 km/h and 10% slope;
* ABI ≥1.00 and ≤1.40.
* Obtained informed consent.

Exclusion Criteria:

Arteriopatic patients :

* Patients with a pacemaker or defibrillator;
* Patients with acute or critical limb ischemia;
* Ambulation limited by exertional symptoms other than intermittent claudication (e.g., dyspnea or angina pectoris);
* Ambulation limited by exertional symptoms indicative of intermittent claudication but affecting muscles in the lower extremities other than the calves;
* Contraindication to exercise testing according to the American Heart Association and the American College of Sports Medicine;
* Major cardiovascular event (myocardial infarction or stroke) or major surgery within the previous three months before inclusion;
* Female patients who are pregnant, planning to become pregnant, or lactating;
* Known presence of an aneurysm of the abdominal aorta > 4cm or an aneurysm of the iliac artery >1.5cm;
* Patient subject to legal protection (guardianship or tutelage measure) and persons deprived from their liberty (according to French law);
* Simultaneous participation to another ongoing clinical research protocol;
* Unwilling or unable to engage in the completion of a 12 week programme;
* Any planned event(s) that could interfere with the completion of the protocol: e.g., extended holidays preventing the completion of the intervention or planned hospitalization for a prolonged period of time.
* Body mass > 160 kg (may exceed treadmill limit).
* Inability to understand and sign informed consent forms due to cognitive or language barriers
* LEPAD due to other causes than atherosclerosis.

Healthy volunteers :

* Contraindication to walking;
* ABI <1.00 or >1.40;
* Inability to obtain a measure of ABI due to uncompressible arteries;
* Limitation(s) and/or symptoms during the treadmill walking test;
* Treadmill walking test uncompleted.
* Presence of hypertension, heart failure, angina pectoris, diabetes, chronic obstructive pulmonary disease, supported by the presence of a medical treatment and the medical history.
* Presence of conditions likely to cause a functional limitation in walking and/or significant modification of physiological responses to the exercise: current or former smoker from less than 6 months, cancer (ongoing), Parkinson's disease, renal failure (ongoing), supported by the presence of a medical treatment and the medical history.
* History of cardiovascular disease (heart failure, stroke, myocardial infarction) reported by the patient.
* Female volunteers who are pregnant, planning to become pregnant, or lactating;
* Volunteers subject to legal protection (guardianship or tutelage measure) and persons deprived from their liberty (according to French law).
* Simultaneous participation to another ongoing clinical research protocol.

Secondary exclusion criteria for patients :

1. Patients requiring a pacemaker or defibrillator within the first three months.
2. For the primary endpoint, patients who underwent revascularisation (surgical or endovascular) in the first three months.

   revascularisation (surgical or endovascular) in the first three months.
3. 3. Any health events during the first three months that no longer allow the patient to follow the protocol.
4. Burning during the electrostimulation sessions;
5. Skin allergy due to the placement of the electro-stimulation electrodes

Min Age: 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Change in treadmill walking distance to maximal leg pain (absolute walking distance) | 12 weeks
  Comparison of change in treadmill walking distance to maximal leg pain (absolute walking distance) after 12 weeks between ESM group and control group (between visit 1 and visit 2)

SECONDARY OUTCOMES:
Change in treadmill walking distance to onset of leg pain | 12 weeks
  Comparison of change in treadmill walking distance to onset of leg pain between visit 1 and visit 2, and between NMES and control group
Change in 6-minute total walk distance | 12 weeks
  Comparison of change in 6-minute total walk distance between visit 1 and visit 2, and between NMES and control group
Change in maximal walking distance and medium walking speed under natural outdoor conditions | 12 weeks
  Comparison of change in maximal walking distance and medium walking speed under natural outdoor conditions between visit 1 and visit 2, and between NMES and control group
Change in the Walking Impairment Questionnaire score | 12 weeks
  Comparison of change in the Walking Impairment Questionnaire (WIQ) score between visit 1 and visit 2 and between NMES and control group. the WIQ is a valid tool to detect improvement or deterioration in the daily walking ability of patients with intermittent claudication. The higher the WIQ score is, the better the patient's functional walking ability is.
Change in the Short Form (36) Health Survey (SF36) score | 12 weeks
  Comparison of change in the Short Form (36) Health Survey (SF36) score between visit 1 and visit 2, and between NMES and control group. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software.
Change in the Peripheral Artery Questionnaire (PAQ) score | 12 weeks
  Comparison of change in the Peripheral Artery Questionnaire score between visit 1 and visit 2, and between NMES and control group. The Peripheral Artery Questionnaire (PAQ) is a 20-item questionnaire developed to meet this need by quantifying patients' physical limitations, symptoms, social function, treatment satisfaction, and quality of life. higher scores represent fewer symptoms and better health status
Change in in actigraphy measures | 12 weeks
  Comparison of change in actigraphy measures to define daily physical activity level between visit 1 and visit 2 and between NMES, and control group
Change in ankle brachial index | 12 weeks
  Comparison of change in ankle brachial index between visit 1 and visit 2, and between NMES and control group. The ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium). Compared to the arm, lower blood pressure in the leg suggests blocked arteries due to peripheral artery disease (PAD). The ABI is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressure in the arm
Change in TcPO2 DROP during treadmill walking test | 12 weeks
  Comparison of change in TcPO2 DROP during treadmill walking test between visit 1 and visit 2 and between NMES and control group
Number of patients submitted to a revascularization procedure | 12 weeks
  Comparison in the number of patients submitted to a revascularization procedure between visit 1 and visit 2, and between NMES and control group
Change in results of Contrast imaging with laser granularity | 12 weeks
  Comparison of change in endothelial function using Contrast imaging with laser granularity, only for arteriopathic patients included in Rennes, between visit 1 and visit 2 and between NMES and control group. Laser Contrast Granularity Analysis is a method that allows the visualization of tissue blood perfusion instantly in real time.
Percentage of physiological response achieved by patients | 12 weeks
  Percentage of physiological response achieved by patients for all outcome measures (comparison with parameters of volunteers without any cardiac or vascular disease) between all visits
Change in maximum walking distance according to the location of the arterial obstruction | 12 weeks
  Change in maximum walking distance according to the location of the arterial obstruction using scan images between visit 1 and visit 2 and between NMES and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mahe, Pr, Principal Investigator — Rennes University Hospital
Locations (5):
- France (5):
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHU de Rennes, Rennes
  - Hôpital de Rangueil, Toulouse

REFERENCES:
- [Derived] Le Faucheur A, Chanteau A, Jehannin P, Le Pabic E, Houssein A, Talbot M, Mimassi ML, Donnelly A, Espinasse B, Lecoq S, Bura-Riviere A, Kaladji A, Laneelle D, Mahe G. Effect of a home-based calf neuromuscular electrical stimulation program on walking capacity in adults with lower-extremity PAD: the ELECTRO-PAD RCT. Eur J Prev Cardiol. 2026 Feb 9:zwag080. doi: 10.1093/eurjpc/zwag080. Online ahead of print. PMID 41662341
- [Derived] Jehannin P, Craughwell M, Omarjee L, Donnelly A, Jaquinandi V, Mahe G, Le Faucheur A. A systematic review of lower extremity electrical stimulation for treatment of walking impairment in peripheral artery disease. Vasc Med. 2020 Aug;25(4):354-363. doi: 10.1177/1358863X20902272. Epub 2020 Apr 17. PMID 32303155